CLINICAL TRIAL: NCT03343990
Title: Comparison Between Interlocking Multi-twisted Wires and Eight Figure of Sternum Closure Post Open Heart Surgery in Egyptian Patients
Brief Title: Comparison Between Interlocking Multi-twisted Wires and Eight Figure of Sternum Closure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Rabee Hamed Ahmed, sternal closure, Assiut University
Other Study IDs: sternal closure
Record Dates: First submitted 2017-09-08; First posted 2017-11-17 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Sternotomy Closure,Open Heart Surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- group A: Interlocking multi-twisted wires techniqe in sternal closure
  Interventions: Procedure: Interlocking multi-twisted wires in sternal closure; Procedure: Eight Figure techniqe in sternal closure
- group B: Eight Figure techniqe in sternal closure
  Interventions: Procedure: Interlocking multi-twisted wires in sternal closure; Procedure: Eight Figure techniqe in sternal closure

INTERVENTIONS:
Procedure: Interlocking multi-twisted wires in sternal closure — One of many ways in cloure of sternal give more stabilization. At least 6 wires have to be passed. The wirs should run around the sternum in the intercostals spaces except in the manubrium where it has to be passed through the bone . Adjacent wires on the surgeon's side are wrapped around each other. The wires on the surgeon's side are then pulled towards the assistant so that the sternum is re-approximated. Alternatively the surgeon can also pull the wires at the assistant's side towards himself or herself approximating the sternum. Adjacent wires on the assistant's side are then wrapped around each other. The wrapped wires on both sides are then wrapped around each other The wrapped wires are then twisted around with a twister, closing the sternum tightly and the ends of the are burried
  Other Names: prakash p.punjabi
Procedure: Eight Figure techniqe in sternal closure — The figure-eight closure is described as faster, simpler, and more reliable than its trans-sternal counterpart; with only oblique forces sutures are less likely to loosen or fracture the sternum. The advantage of figure-eight closure is that it allows oblique and horizontal angle of shearing forces instead of direct perpendicular forces. Thus these wires are less likely to loosen or fracture

SUMMARY:
Comparison between interlocking multi-twisted wires and Eight figure of sternum closure post open heart surgery in egptian patients

DETAILED DESCRIPTION:
Comparison between interlocking multi-twisted wires and Eight figure of sternum closure post open heart surgery in egptian patients

Midline sternotomy, first described by Milton in 1887 [4,7,8] remains the most popular technique of cardiac exposure because of its quick and easy performance, excellent access to the heart and great vessels. Effective prevention methods for disruption and infection of median sternotomy continue to be debated. The most important factor in preventing PSWC is a stable sternal approximation, as bony union depends on adequate reduction and immobilization of the stern costal junctions. Strict adherence of preoperative aseptic technique is crucial. Careful attention to homeostasis and meticulous surgical technique remain the mainstays of prevention and must include precise sternal alignment and stable closure. While biomechanical studies appear to be valid, their general value is limited Different sternal closure techniques

1. Trans-sternal/peristernal wiring
2. Bilateral and longitudinal parasternal running wires (described by Robicsek)
3. Double wires
4. Steel band
5. Figure of eight The figure-eight closure is described as faster, simpler, and more reliable than its trans-sternal counterpart; with only oblique forces sutures are less likely to loosen or fracture the sternum. The advantage of figure-eight closure is that it allows oblique and horizontal angle of shearing forces instead of direct perpendicular forces. Thus these wires are less likely to loosen or fracture .
6. Interlocking multi-twisted wires One of recent way in closure of sternal gives more stabilization. At least 6 wires have to be passed. The wires should run around the sternum in the intercostals spaces except in the manubrium where it has to be passed through the bone . Adjacent wires on the surgeon's side are wrapped around each other. The wires on the surgeon's side are then pulled towards the assistant so that the sternum is re-approximated. Alternatively the surgeon can also pull the wires at the assistant's side towards himself or herself approximating the sternum. Adjacent wires on the assistant's side are then wrapped around each other. The wrapped wires on both sides are then wrapped around each other the wrapped wires are then twisted around with a twister, closing the sternum tightly and the ends buried

6- Alternative techniques

Techniques utilizing lateral sternal support are first-line options in preventing SD and wound infections. The need to provide lateral reinforcement of the sternum has led to the development of several techniques, such as A-the use of lateral staples and lateral plates B-H-shaped titanium plates C- Reinforced sternal closure system D-thermo reactive clips E- Rigid plate fixation change

The purpose of this report was to analyze (I) the efficacy of most used ways in sternal closure in our center ( interlocking multi-twisted wires and Eight figure )for the prevention of Post sternal wound complication in adult egyptian patients and find the way more efficient in sternal closure.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient above 16 years undergoing open heart surgery with sternotomy
2. Patient is willing to comply with all follow-up visits.
3. Willing and able to provide written informed consent and comply with study requirements

Exclusion Criteria:

1. Pediatric patients below 16 years
2. Extra-cardiac illness that is expected to limit survival to less than 5 years e.g. oxygen-dependent chronic obstructive pulmonary disease, active hepatitis or significant hepatic failure, severe renal disease.

Ages: 17 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adult patient above 16 years undergoing open heart surgery with sternotomy
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2019-03-29 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Healing of the sternum | 60 days
  Duration of complete healing of the sternum :By
  1. Radiological (chest x-ray ant-post view and lat view in first 6 weeks post-operative
  2. Clinical examination in first 6 weeks post operative

SECONDARY OUTCOMES:
rate of wound infection | 30 days
  way less liable to infect wound either skin infection or wound dehiscence
mobilization | 45 days
  Early mobilization after surgery till returning to normal movement including freely arm movement
Time of procedure | 45 days
  time taken by each way in sternal closure

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Information collected by this study may contribute to decrease postoperative complication as sternal dehescince , improve local wound complication & decrease cost by decrease hospital stay & need for antibiotics needed for wound infection and rewiring. On the other hand patients will benefit from the clinical and radiological follow up postoperatively. There are no known risks associated with participation in this study. Patients' treatment and follow up will not be altered by any means.

REFERENCES:
- [Result] Karra R, McDermott L, Connelly S, Smith P, Sexton DJ, Kaye KS. Risk factors for 1-year mortality after postoperative mediastinitis. J Thorac Cardiovasc Surg. 2006 Sep;132(3):537-43. doi: 10.1016/j.jtcvs.2006.04.037. PMID 16935107
- [Result] Song DH, Lohman RF, Renucci JD, Jeevanandam V, Raman J. Primary sternal plating in high-risk patients prevents mediastinitis. Eur J Cardiothorac Surg. 2004 Aug;26(2):367-72. doi: 10.1016/j.ejcts.2004.04.038. PMID 15296898
- [Result] Bottio T, Rizzoli G, Vida V, Casarotto D, Gerosa G. Double crisscross sternal wiring and chest wound infections: a prospective randomized study. J Thorac Cardiovasc Surg. 2003 Nov;126(5):1352-6. doi: 10.1016/s0022-5223(03)00945-0. PMID 14666006
- [Result] Losanoff JE, Collier AD, Wagner-Mann CC, Richman BW, Huff H, Hsieh Fh, Diaz-Arias A, Jones JW. Biomechanical comparison of median sternotomy closures. Ann Thorac Surg. 2004 Jan;77(1):203-9. doi: 10.1016/s0003-4975(03)01468-1. PMID 14726062
- [Result] Robicsek F, Fokin A, Cook J, Bhatia D. Sternal instability after midline sternotomy. Thorac Cardiovasc Surg. 2000 Feb;48(1):1-8. doi: 10.1055/s-2000-9945. PMID 10757149
- [Result] Schimmer C, Sommer SP, Bensch M, Leyh R. Primary treatment of deep sternal wound infection after cardiac surgery: a survey of German heart surgery centers. Interact Cardiovasc Thorac Surg. 2007 Dec;6(6):708-11. doi: 10.1510/icvts.2007.164004. Epub 2007 Sep 20. PMID 17884847
- [Result] Noyez L, van Druten JA, Mulder J, Schroen AM, Skotnicki SH, Brouwer RM. Sternal wound complications after primary isolated myocardial revascularization: the importance of the post-operative variables. Eur J Cardiothorac Surg. 2001 Apr;19(4):471-6. doi: 10.1016/s1010-7940(01)00610-8. PMID 11306315
- [Result] [11] Prakash.P.Punjabi Essentials_of_Operative cardiac surgery page 62 chest closure